CLINICAL TRIAL: NCT00174161
Title: The Symptom Experience of Women With Perimenstrual Syndrome;Women's Health Related Quality of Life.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700617; NSC93-2314-B002-054; NSC94-2314-B002-009
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome,Health Related Quality of Life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Self Care

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: self-care, health behavior

SUMMARY:
The purpose of these series research project is to investigate the prevalence, symptoms cluster and characteristic; establish the systemic symptom management nursing strategies (PMS-SMP); determine short-and long-term effectiveness of PMS-SMP. To enhance the health related quality of life of women with Perimenstrual syndrome. Simultaneously, the PMS-SMP offers a research and clinical based protocol to demonstrate the independent nursing role and practice care model. The 3-year series research process will include three research domains.

DETAILED DESCRIPTION:
Symptoms are the most common reason people seek health care. Although the menstrual cycle, a normative process, but 10~15% of western women experience sever recurring symptoms associated with the menstrual cycle that can be considered a chronic illness. There are many interventional researches focus on this issue in western countries. There is not only lack of evidence base prevalence of perimenstrual syndrome, but also never found any nursing intervention project focusing on women with perimenstrual syndrome.

The purpose of these series research project is to investigate the prevalence, symptoms cluster and characteristic; establish the systemic symptom management nursing strategies (PMS-SMP); determine short-and long-term effectiveness of PMS-SMP. To enhance the health related quality of life of women with Perimenstrual syndrome. Simultaneously, the PMS-SMP offers a research and clinical based protocol to demonstrate the independent nursing role and practice care model. The 3-year series research process will include three research domains.

Content analysis, descriptive statistics(percentage, mode, medium, quartile, rank), Chi-square, One way ANOVA, MANCOVA, and Step-Wise regression will be applied to examine the research finding. Although focused on perimenstrual symptoms relief and improve the health related quality of life of women with perimenstrual symptoms, these strategies are generally health promoting and can be applied to other women's health conditions.

ELIGIBILITY:
Inclusion Criteria:

* female

Exclusion Criteria:

* pregnancy,menopause,woman with breast-feeding

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-08; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Yang Ya Ling, Study Chair — National Taiwan University Hospital
Locations (1):
- NTUH, National Taiwan University Hosptal, Taipei, 7, Chung-Shan South Road, Taiwan